CLINICAL TRIAL: NCT05778071
Title: A Phase 3 Multicenter, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Efficacy and Safety of Eneboparatide (AZP-3601), a Parathyroid Hormone Receptor Agonist, in Patients With Chronic Hypoparathyroidism (CALYPSO)
Brief Title: Evaluation of the Safety and Efficacy of Eneboparatide (AZP-3601) in Patients With Chronic Hypoparathyroidism
Acronym: CALYPSO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Amolyt Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZP-3601-CLI-002
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hypoparathyroidism; Endocrine System Diseases; Parathyroid Diseases
Keywords: Hypoparathyroidism
MeSH Terms: conditions — Endocrine System Diseases; Parathyroid Diseases; Hypoparathyroidism

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind study, with patients randomized in a 2:1 ratio to receive eneboparatide or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- eneboparatide (Experimental): Starting dose of 20 mcg; Administered once daily by subcutaneous injection
  Interventions: Combination Product: eneboparatide
- Placebo (Placebo Comparator): Administered once daily by subcutaneous injection
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: eneboparatide — Supplied as a solution (concentration of 250 mcg/mL or 500 mcg/mL) in single-patient-use prefilled pens
  Other Names: AZP-3601
  Arms: eneboparatide
Combination Product: Placebo — Placebo is supplied as a solution (containing the excipient solution for eneboparatide) in single-patient-use prefilled pens
  Arms: Placebo

SUMMARY:
This study is investigating the safety and efficacy of eneboparatide (AZP-3601) in patients with chronic hypoparathyroidism (cHP).

During the first 24 weeks of the trial, participants will be randomized to receive eneboparatide or placebo. Study treatment is blinded: patients and doctors will not know which group each patient has been randomized to. All patients will start with a fixed dose of study treatment (eneboparatide or placebo), administered subcutaneously with a pre-filled pen. Study treatment will be individually titrated.

After completion of the first 24 weeks, patients will be treated in the open label extension part of the study for 132 weeks. During this phase, all patients (including patients that were in the placebo group) will receive eneboparatide.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females, 18-80 years of age
2. Patients with cHP for ≥12 months at the time of screening
3. Two paired measurements of showing low parathyroid hormone (PTH) and serum calcium either below normal or within normal under standard of care
4. Requirement for therapy with calcitriol ≥0.5 mcg per day or alphacalcidol ≥1 mcg per day, and requirement for supplemental oral calcium treatment ≥1000 mg per day over and above patient's dietary calcium intake at Day 1 visit
5. Successful completion of the Optimization period based on two consecutive measurements of albumin-adjusted serum calcium at least 1 week apart within the range of 7.8 to 9.0 mg/dL and with no more than 25% of change in the daily dose of any of active vitamin D and oral calcium supplements between the two measurements
6. Thyroid-stimulating hormone (TSH) within the lower limit of normal and 1.5-fold of the upper limit of normal at screening; if on suppressive therapy for a history of thyroid cancer, TSH level must be ≥0.2 mIU/mL and thyroid medication should be stable for at least 6 weeks prior to treatment
7. Prior to start of treatment:

   * Magnesium level within laboratory normal limits
   * 25(OH) vitamin D levels of 30-70 ng/mL (75-175 nmol/L)
8. eGFR ≥30 mL/min/1.73m² during screening
9. Able to perform daily subcutaneous self-injections of study drug (or have a designee to perform injections) via a pre-filled injection pen
10. Female patients of non-childbearing potential or using an effective method of contraception throughout the study. Women of childbearing potential should have a negative pregnancy test.
11. Able and willing to provide written and signed informed consent in accordance with GCP

Exclusion Criteria:

1. Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation
2. Clinically significant abnormal values at screening for hematology, clinical chemistry, coagulation or urinalysis
3. Abnormal arterial pressure at screening, defined as (1) systolic blood pressure <100 mmHg, or (2) systolic blood pressure >150 mmHg, and/or diastolic blood pressure >100 mmHg.
4. Heart rate at rest outside the range of 50-100 beats/minute at screening
5. Clinically significant abnormal standard 12-lead electrocardiogram indicative of severe cardiac disease
6. Known history of autosomal-dominant hypocalcemia or known pseudohypoparathyroidism (impaired responsiveness to PTH)
7. Any current disease (other than hypoparathyroidism) that might affect calcium metabolism, calcium-phosphate homeostasis or PTH levels
8. Patients with increased risk for osteosarcoma
9. Current uncontrolled active disease processes that may adversely affect gastrointestinal absorption
10. History of cerebrovascular accident within 6 months prior to screening
11. History of active uncontrolled malignancy over the past 2 years at time of screening
12. History of any other cancer other than thyroid cancer (except basal cell skin cancer or squamous cell skin cancer) who have not been disease-free for a period of at least 2 years at the time of screening
13. Acute gout <2 months prior to screening
14. Dependent on parenteral calcium infusions to maintain calcium homeostasis
15. Use of medications such as loop and thiazide diuretics, raloxifene hydrochloride, lithium, methotrexate, cardiac glycosides or systemic corticosteroids within 4 weeks prior to start of treatment
16. Previous treatment with PTH/parathyroid hormone-related protein-like drugs, including PTH(1-84) and PTH(1-34) within 3 months of screening
17. Use of other drugs known to influence calcium and bone metabolism within 4 weeks of screening
18. Use of oral bisphosphonates within 6 months of screening or intravenous bisphosphonate within 12 months of screening
19. Use of denosumab within 18 months of screening
20. Seizure disorder/epilepsy with history of a seizure within 6 months of screening
21. History of symptomatic urinary tract calculi within 3 months of screening
22. Irradiation to the skeleton within 2 years of screening
23. Pregnant or breastfeeding female patients
24. Participation in any other interventional study in which the patient received an investigational drug or device within 2 months or within 5 times the half-life of the investigational drug (whichever comes first) prior to screening
25. Any disease or condition that, in the opinion of the investigator, may require treatment or make the subject unlikely to fully complete the trial, or any condition that presents undue risk from the study treatment or procedures, including treated malignancies that are likely to recur within the approximate duration of the trial
26. Any other reason that in the opinion of the investigator would prevent the subject from completing participation or following the trial schedule
27. Known allergy or sensitivity to PTH or any of the excipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2027-06-16 (Estimated)

PRIMARY OUTCOMES:
Efficacy - Primary Endpoint | 24 weeks
  After 24 weeks of treatment, the proportion of patients in the eneboparatide treatment group vs. placebo:
  * Achieving complete independence from active vitamin D;
  * Achieving independence from therapeutic doses of oral calcium (i.e. taking oral elemental calcium supplements ≤600 mg/day); and
  * With albumin-adjusted serum calcium within the normal range (8.3 to 10.6 mg/dL).

SECONDARY OUTCOMES:
Hypercalciuria | 24 weeks
  Proportion of patients who had hypercalciuria at baseline and normalize 24-hour urinary calcium excretion level (i.e., achieve <250 mg/24 hours for females or <300 mg/24 hours for males)
Change from baseline in the HPT-DD-SE - Physical Domain score | 24 weeks
  Change from baseline in patient's symptoms, as assessed by the average weekly HPT-DD-SE physical domain score in the eneboparatide treatment group vs. placebo
Change from baseline in the HPT-DD-SE - Cognitive Domain score | 24 weeks
  Change from baseline in patient's symptoms, as assessed by the average weekly HPT-DD-SE cognitive domain score in the eneboparatide treatment group vs. placebo
Change from baseline in the HPT-LIQ - Physical Functioning Domain score | 24 weeks
  Change from baseline in the HPT-LIQ Physical Functioning domain score, in the eneboparatide treatment group vs. placebo
Change from baseline in the SF-36 Physical Functioning subscore | 24 weeks
  Change from baseline in the SF-36 Physical Functioning subscore in the eneboparatide treatment group vs. placebo

CONTACTS AND LOCATIONS:
Overall Officials: Soraya Allas, MD, Study Director — Amolyt Pharma
Locations (54):
- United States (16):
  - Harbor UCLA Medical Center Endocrinology, Torrance, California
  - Denver Endocrinology Diabetes and Thyroid Center, Denver, Colorado
  - University of Chicago - Medical Center, Chicago, Illinois
  - North Shore University Health System, Evanston, Illinois
  - Indiana University (IU) Health University Hospital, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Northern Nevada Endocrinology, Reno, Nevada
  - Colombia University Irving Medical Center, New York, New York
  - Physician's East Endocrinology, Greenville, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - The Children's Hospital of Philadephia, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Academy of Diabetes, Thyroid and Endocrine, El Paso, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
- Canada (3):
  - Eastern Regional Health Authority Health Sciences Centre, St. John's, Newfoundland and Labrador
  - Bone Research and Education Center, Oakville, Ontario
  - CHU de Quebec Research Centre, Québec
- Denmark (2):
  - Aarhaus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (3):
  - Hopital de la Conception-APHM, Marseille
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - Hospital Bicetre AP-HP, Paris
- Germany (3):
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Medicover Neuroendokrinologie MVZ, Munich
  - Universitaetsklinikum Wuerzburg, Würzburg
- Hungary (2):
  - Semmelweis Egyetem Belgyogyaszati es Hematologiai Klinika, Budapest
  - Pecsi Tudomanyegyetem, Pécs
- Italy (5):
  - Azienda Ospedaliero Universitaria de Bologna, Policlinico Sant Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Azienda Ospedaliera Universitaria Pisana-Ospedale di Cisanello, Pisa
  - Via Alvaro del Portillo, 200, Roma, Italy 00128, Roma
- Japan (6):
  - Teikyo University Chiba Medical Center, Chiba
  - Kanazawa University Hospital, Kanazawa
  - Osaka City Hospital, Osaka
  - Osaka Metropolital University Hospital, Osaka
  - Tokushima University Hospital, Tokushima
  - Tottori University Hospital, Tottori
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Eramus MC - University Medical Center, Rotterdam
- Poland (3):
  - Medycyny Nuklearnej i Chorob Wewnetrznych, Krakow
  - Instytut Centrum Zdrowia Matki Polki. Klinika Endokrynologii Chorob Metabolicznych, Lodz
  - Cendrum Zdrowi MDM - EB Group Sp., Warsaw
- Portugal (2):
  - Hospital da Luz Lisboa, Lisbon
  - Centro Hospital Vila Nova de Faia/Espinho, Porto
- Spain (4):
  - Complejo Hospitalario Universitario de A Coruna, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (3):
  - University Hospitals of Leicester NHS Trust, Leicester
  - Norfolk & Norwich University NHS Foundation Trust, Quadrum Institute, Norwich
  - Churchill Hospital, Oxford